CLINICAL TRIAL: NCT01733303
Title: Fracture and Fall Prevention in Elderly With Osteoporosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 201003065R
Record Dates: First submitted 2012-10-05; First posted 2012-11-27 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (1):
- Exercise (Experimental): Participants are allocated to the exercise group will commence the personalized core training exercise with EMG biofeedback based on their testing results in muscle quality.
  Interventions: Behavioral: personalized core muscle training program

INTERVENTIONS:
Behavioral: personalized core muscle training program — Participants are allocated to the exercise group will commence the personalized core training exercise with EMG biofeedback based on their testing results in muscle quality. The program will run for 3 months with patients attending for one hour three times a week. The age-matched control group will maintain their usual daily life activities without any specific instruction. The exercise training will be run by an experienced physiotherapist, who will encourage patients individually to progress at their own pace.

SUMMARY:
Osteoporosis is a prevalent health concern among older adults and is associated with an increased risk of falls that can cause fracture, injury or mortality. Identifying the factors related to falls occurring within this population is essential for the development of effective regimes for fall prevention. Studies have shown that muscle quality and good posture alignments are critical for balance control in older adults. People are diagnosed with osteoporosis often combining with muscles weakness, and increased spine kyphosis leading vertebral, fractures and poor balance control, even falls. Therefore, improving muscle quality, strengthening weak muscles and correcting postural alignment are essential elements for fracture and fall prevention in older adults with osteoporosis. The long-term objectives of this work are to prevent fracture and fall in older adults with osteoporosis by improving the function of degenerative muscles using exercise training.

ELIGIBILITY:
The inclusion criteria for osteopenia or osteoporosis group:

1. able to stand and walk for 5 minutes independently;
2. having normal or corrected to normal vision;
3. having age between > 50 years
4. with osteopenia (-2.5 < t-score < -1.0) or osteoporosis (t-score <-2.5).

The exclusion criteria for osteopenia or osteoporosis group:

1. being pregnant;
2. sensory-motor deficits;
3. inability of communication
4. lack of access to a telephone.

The inclusion criteria for control age-matched group:

1. able to stand and walk for 5 minutes independently;
2. having normal or corrected to normal vision;
3. having age between > 50 years
4. without osteopenia or osteoporosis (t-score > -1.0).

The exclusion criteria for control age-matched group:

1. being pregnant;
2. sensory-motor deficits;
3. inability of communication
4. lack of access to a telephone.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Changes of torque demand to capacity ratio 6 months | Change from Baseline intorque demand to capacity ratio at 6 months
Changes of torque demand to capacity ratio at 3 months | Change from Baseline in torque demand to capacity ratio at 3 months
Change of torque demand to capacity ratio at 12months | Change from Baseline in torque demand to capacity ratio at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Weili Hsu, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Physical Therapy Center or the Orthopedic Center in the National Taiwan University Hospital, Taipei, Taiwan, Taiwan